CLINICAL TRIAL: NCT03656133
Title: Use of a Proliferation Saturation Index to Determine Personalized Radiotherapy Fractionation for Patients With HPV+ Oropharyngeal Cancers
Brief Title: Use of a Proliferation Saturation Index to Determine Personalized Radiotherapy for HPV + Oropharyngeal Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19579
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Oropharyngeal Cancer
Keywords: HPV; Radiotherapy Fractionation; Proliferation Saturation Index; Larynx; Pharynx
MeSH Terms: conditions — Oropharyngeal Neoplasms; Laryngeal Diseases | interventions — Chemical Fractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Fractionation (Experimental): Investigators will use an individual patient proliferation saturation index (PSI) to select radiotherapy fractionation (conventional fractionation or hyperfractionation) to improve the likelihood of a rapid response (defined as ≥ 32% reduction in volume at 4 weeks).
  Radiotherapy fractionation: Standard fractionation at 2Gy once daily or Hyperfractionation at 1.2 Gy twice daily (≥ 6 hours apart)
  Interventions: Radiation: Radiotherapy fractionation

INTERVENTIONS:
Radiation: Radiotherapy fractionation — Standard fractionation at 2Gy once daily or Hyperfractionation at 1.2 Gy twice daily (≥ 6 hours apart)

SUMMARY:
This study is to determine whether a mathematical model can be used to choose a radiation delivery method to improve the rate of a rapid response.

DETAILED DESCRIPTION:
Investigators hypothesize that using individual patient proliferation saturation index (PSI) to select radiotherapy fractionation (conventional fractionation or hyperfractionation) may improve the likelihood of a rapid response (defined as ≥ 32% reduction in volume at 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥ 18 years
* Pathologically (histologically or cytologically) proven diagnosis of p16+ or HPV+ squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma) of the oropharynx; cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx. Clinical evidence should be documented, and may consist of pathology, palpation, imaging, or endoscopic evaluation, and should be sufficient to estimate the size of the primary (for T stage).
* American Joint Committee on Cancer (AJCC) 8th edition staging T1-3 N0-1 MO
* Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations.
* CT or MRI performed at least 1 week apart. This can consist of diagnostic imaging and radiation therapy planning imaging.
* No evidence of distant metastases
* Eastern Cooperative Oncology Group Performance Status 0 to 3

Exclusion Criteria:

* Age < 18
* Positive urine pregnancy test
* Evidence of distant metastases
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that remove all clinically and radiographically evident disease
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patients with a medical condition or social situation that at the discretion of the PI would preclude them from completion of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Caudell, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiotherapy Fractionation
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy Fractionation
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Response at Week 4 of Treatment
Description: Fractionation of radiation will be individualized based on patient Proliferation Saturation Index (PSI). Objective is to increase the rate of response of ≥ 32% at 4 weeks to 63% of patients, above the expected 49%. Result is reported as percentage of participants who met the criteria for ≥ 32% reduction in tumor volume by week 4.
Time Frame: At 4 weeks of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Radiotherapy Fractionation
Number analyzed (Participants) | 55
percentage of participants | 61.2

2. Secondary Outcome: Rate of Complete Response at 2-3 Months
Description: Rate of complete response by Computed Tomography (CT) at 2 months or Positron Emission Topography (PET)/CT at 3 months following completion of therapy
Time Frame: 2-3 months post treatment
Population: Evaluable participants at 2-3 months post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Radiotherapy Fractionation
Number analyzed (Participants) | 53
percentage of participants
  Complete anatomic and/or metabolic response | 98.1
  Partial anatomic and/or metabolic response | 2.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date participant signed informed consent to 7 days for non serious or 30 days for serious adverse events after last day of study participation, an average of 1 year.
Arm/Group | Radiotherapy Fractionation
All-Cause Mortality (participants affected / at risk) | 2/55
Serious Adverse Events (participants affected / at risk) | 1/55
Other Adverse Events (participants affected / at risk) | 7/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy Fractionation (N=55)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy Fractionation (N=55)
Mucositis oral (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (4)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT03656133/Prot_SAP_000.pdf